CLINICAL TRIAL: NCT07401043
Title: Effects of Solution-Focused Approach on Mothers Anxiety About Preterm Infants Care
Brief Title: Mothers Anxiety About Preterm Infants Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurcan Akgül Gündoğdu (Other)
Responsible Party: Sponsor-Investigator, Nurcan Akgül Gündoğdu, Associate Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BANÜ-SBF-NAG-01
Record Dates: First submitted 2025-12-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Maternal Anxiety
Keywords: Mother having a preterm infant; Preterm infants care; Anxiety level; Solution-Focused Approach; Nursing

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Single-blind: Participants did not know their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solution-Focused Approach (SFA) (Experimental): Mothers in this arm received an Individual Solution-Focused Approach (SFA) intervention consisting of eight 30-45-minute sessions. Three sessions were conducted in the mother-infant harmony room during the NICU discharge process and five sessions were conducted at home during scheduled home visits. SFA techniques included goal setting, identifying exceptions, miracle questions, scaling, reframing, and letter writing. The intervention aimed to reduce maternal anxiety related to caring for a preterm infant and to improve solution-focused thinking skills.
  Interventions: Behavioral: Solution-Focused Approach (SFA)
- Standard Care Control (No Intervention): Mothers in this arm received routine NICU discharge education and standard postpartum care as provided by the hospitals. No additional psychological or behavioral intervention was given between the pre-test and follow-up assessments. After the study was completed, SFA sessions were offered to mothers in the control group.

INTERVENTIONS:
Behavioral: Solution-Focused Approach (SFA) — The intervention consisted of eight individual Solution-Focused Approach (SFA) sessions lasting 30-45 minutes each. Three sessions were provided in the NICU mother-infant harmony room during the discharge process and five sessions were conducted at home during planned home visits. Techniques included goal setting, identifying exceptions, miracle questions, scaling, reframing, and letter writing. The intervention aimed to reduce maternal anxiety related to caring for a preterm infant and to improve solution-focused thinking skills.
  Arms: Solution-Focused Approach (SFA)

SUMMARY:
It has been reported that mothers of preterm infants who experience anxiety face challenges in participating in infant care. However, the effect of solution-focused approach on reducing the anxiety of mothers of premature infants is unknown. This study was conducted to assess the effects of Solution-Focused Approach on the anxiety levels of mothers who are anxious about preterm infants care. A randomized controlled trial design. The present study was carried out in the Neonatal Intensive Care Units of three hospitals in a city center. In the study, the sample group was determined as 40 mothers, 20 of whom were interventions and 20 were control. In this study, eight 30-40minute solution-focused interviews were held with the participants in the intervention group subjected to the Solution Focused Approach. Of the mothers in the intervention group, 5% had triplet pregnancy, 75% gave birth by cesarean section, 80% had health problems during pregnancy and 95% did not receive training on infant care during pregnancy. The differences in scale scores obtained during follow-ups were greater in the intervention group than in the control group. It was determined that the intervention undergone by the mothers of the preterm infants in the intervention group decreased the mothers' anxiety levels about infant care and increased their solution-focused coping skills. Following the intervention, moms in the intervention group showed improvement in all of their self-perception skills about their care needs. The Solution-Focused Approach decreased state-trait anxiety levels of mothers who were anxious about preterm infant care, and improved their solution-focused coping skills. The Individual Solution-Focused Approach decreased state and trait anxiety levels of primiparous mothers who were anxious about preterm infant care, and improved their solution-focused coping skills. Nurses' application of this approach can reduce the anxiety levels of mothers who are worried about preterm infant care. It can contribute to mothers to develop a solution-focused perspective.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mothers
* Having a preterm infant hospitalized in the NICU
* Being in the discharge or mother-infant harmony process
* Scoring ≥20 on at least one anxiety inventory
* Ability to communicate in Turkish
* Voluntary participation and written informed consent

Exclusion Criteria:

* Having a serious medical or psychiatric condition preventing participation
* Mother reporting she cannot continue the interviews
* Mother being out of the province during the intervention dates

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
State Anxiety Score | At baseline; one week after completion of the intervention; 2-month after completion of the intervention
  Change in mothers' state anxiety levels measured using the State Anxiety Inventory (20-80 points; higher scores indicate greater anxiety). The scale was administered at baseline; one week after completion of the intervention; 2-month after completion of the intervention.
Trait Anxiety Score | At baseline; one week after completion of the intervention; 2-month after completion of the intervention
  Change in mothers' trait anxiety levels measured with the Trait Anxiety Inventory (20-80 points). Higher scores indicate higher trait anxiety. Measurements were taken at baseline; one week after completion of the intervention; 2-month after completion of the intervention.

SECONDARY OUTCOMES:
Solution-Focused Thinking Skills Score | At baseline; one week after completion of the intervention; 2-month after completion of the intervention
  Change in mothers' solution-focused thinking skills as measured by the Solution-Focused Inventory (12-72 points; higher scores indicate stronger solution-focused thinking). Scale administered at baseline; one week after completion of the intervention; 2-month after completion of the intervention.
Home Care Needs Competence | At baseline; one week after completion of the intervention
  Change in mothers' competencies in providing home care to their preterm infants, measured using the Home Care Needs Evaluation Form for Mothers of Preterm Infants. This form assesses maternal competence across multiple care domains. Higher scores indicate greater competence.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan AKGUL GUNDOGDU, PhD, Assoc. Prof., Principal Investigator — Bandirma Onyedi Eylül University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Sivas Cumhuriyet University Research and Training Hospital - Neonatal Intensive Care Unit (NICU), Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive clinical and psychological information related to mothers and their preterm infants. Although all analyses were conducted using aggregated and de-identified data, the release of raw IPD is not planned due to ethical considerations, confidentiality requirements, and institutional data protection policies.